CLINICAL TRIAL: NCT00870792
Title: Physician Focused Intervention to Improve Adherence With HIV Antiretrovirals
Acronym: MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Ira B. Wilson, MD, MSc, Tufte Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ibwadhrct88$
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2009-03

CONDITIONS: HIV Infection; HIV Infections
Keywords: HIV; antiretroviral therapy; medication adherence; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Received report (Active Comparator)
  Interventions: Behavioral: Adherence report
- Routine care (Placebo Comparator): Patients receive usual, routine, care.
  Interventions: Behavioral: Adherence report

INTERVENTIONS:
Behavioral: Adherence report — During the intervention phase, the data collected at the study visit were summarized in a 3-page report that was given to the provider before each intervention visit. The report included data on self-reported adherence, MEMS adherence, reminder use, beliefs about ART, reasons for missed doses, alcohol and drug use, and depression.

SUMMARY:
We hypothesized that providing physicians treating with HIV disease, at the time of a routine outpatient visit, with a detailed report describing patients' adherence with HIV antiretroviral medications, would improve the quality of the physician-patient interaction, and also patients' subsequent adherence.

ELIGIBILITY:
Inclusion Criteria:

* on ART
* willing to use MEMS cap
* speaks and reads English
* detectable viral loads

Exclusion Criteria:

* uses a pill box

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2002-11; Primary Completion 2005-01 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Antiretroviral medication adherence as assessed by electronic pill cap monitoring. | 6 months

SECONDARY OUTCOMES:
Self-reported medication adherence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ira B. Wilson, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav. 2008 Jan;12(1):86-94. doi: 10.1007/s10461-007-9261-4. Epub 2007 Jun 19. PMID 17577653
- [Background] Vranceanu AM, Safren S, Cowan J, Ring D. The development of the negative pain thoughts questionnaire. Pain Pract. 2008 Sep-Oct;8(5):337-41. doi: 10.1111/j.1533-2500.2008.00213.x. Epub 2008 May 23. PMID 18503620